CLINICAL TRIAL: NCT06731023
Title: Efficacy of a 14-Day Bismuth-Containing Quadruple Therapy Guided by Drug Susceptibility Testing in Patients with Extremely Refractory Helicobacter Pylori Infection: an Exploratory Study
Status: Not yet recruiting | Type: Observational
Sponsor: Xiuli Zuo (Other)
Responsible Party: Sponsor-Investigator, Xiuli Zuo, Professor, Director of gastroenterology department of Qilu hospital., Shandong University
Organization: Shandong University (Other)
Other Study IDs: KYLL-202410-006-1
Record Dates: First submitted 2024-12-08; First posted 2024-12-12 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: HELICOBACTER PYLORI INFECTIONS
Keywords: Helicobacter pylori; Bismuth-Containing Quadruple Therapy; Drug Susceptibility Testing
MeSH Terms: interventions — Bismuth; 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Amoxicillin; Rifabutin; Metronidazole

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Gastric mucosa samples, stool samples, and breath samples obtained during the study will be stored in a specific storage location for 10 years after the study is completed, and then completely deleted after 10 years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Unsuccessful culture attempts group: Bismuth-containing quadruple therapy (vonoprazan 20 mg bid + bismuth 0.6g bid + amoxicillin 1g bid + rifabutin 0.15g bid)
  Interventions: Drug: Bismuth; Drug: Vonoprazan; Drug: Amoxicillin; Drug: Rifabutin
- Demonstrate sensitivity to both amoxicillin and rifabutin group: Bismuth-containing quadruple therapy (vonoprazan 20 mg bid + bismuth 0.6g bid + amoxicillin 1g bid + rifabutin 0.15g bid)
  Interventions: Drug: Bismuth; Drug: Vonoprazan; Drug: Amoxicillin; Drug: Rifabutin
- Drug susceptibility testing group: Two non-resistant antibiotics are selected based on drug susceptibility testing outcomes. If a patient shows sensitivity to only one antibiotic, a combination of that sensitive antibiotic with high-dose metronidazole is administered.
  Interventions: Drug: Bismuth; Drug: Vonoprazan; Drug: Amoxicillin; Drug: Rifabutin; Drug: Metronidazole; Drug: Other antibiotics

INTERVENTIONS:
Drug: Bismuth — Bismuth 0.6g bid
Drug: Vonoprazan — vonoprazan 20mg bid
Drug: Amoxicillin — Amoxicillin 1g bid
Drug: Rifabutin — Rifabutin 0.15g bid
Drug: Metronidazole — Metronidazole 400mg qid
  Groups: Drug susceptibility testing group
Drug: Other antibiotics — The selection of other antibiotics is based on the results of drug susceptibility testing.
  Groups: Drug susceptibility testing group

SUMMARY:
Helicobacter pylori (H. pylori) infection, a prevalent global infectious disease, is a significant contributor to gastric cancer and other morbidities, imposing a substantial disease burden. With the rise in antibiotic resistance, the eradication of H. pylori is encountering formidable challenges. A subset of individuals, despite undergoing multiple treatment regimens, remain unable to successfully eradicate the infection. The persistence of infection in these cases could be attributed to either the limitations of detection methods leading to false positives or to the infection by superbugs that are highly resistant to antibiotics. This study is designed to ascertain whether these patients are infected with superbugs by employing various diagnostic techniques. Additionally, it aims to assess the antibiotic resistance profiles of strains associated with extremely refractory H. pylori infections through drug susceptibility testing. Based on the identified sensitivities, the study seeks to tailor treatment protocols with bismuth-containing quadruple therapy (Containing two kinds of antibiotics: sensitive antibiotic, rifabutin or high-dose metronidazole), to explore novel therapeutic strategies for patients with highly resistant H. pylori infections.

DETAILED DESCRIPTION:
The study enrolled patients with extremely refractory Helicobacter pylori (H. pylori) infection, identified in the outpatient department. Following enrollment, a comprehensive diagnostic approach was employed to ascertain the presence of H. pylori infection and to rule out false positives. Patients who test truly positive for H. pylori should undergo eradication therapy, avoiding any previously administered regimens. For those with unsuccessful culture attempts, a bismuth-containing quadruple therapy (vonoprazan + bismuth + amoxicillin + rifabutin) is recommended as an exploratory approach. Patients with successful cultures should undergo drug susceptibility testing to identify antibiotic resistance patterns of the H. pylori strain. Based on these results, a 14-day course of bismuth-containing quadruple eradication therapy is prescribed. Patients with strains that demonstrate sensitivity to both amoxicillin and rifabutin are assigned to the bismuth-containing quadruple therapy group (vonoprazan + bismuth + amoxicillin + rifabutin). For other patients, two non-resistant antibiotics are selected based on drug susceptibility test outcomes. If a patient shows sensitivity to only one antibiotic, a combination of that sensitive antibiotic with high-dose metronidazole is administered. After eradication treatment, 13C urea breath test and fecal antigen detection were re-examined 4 weeks after drug withdrawal.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-65.
2. Patients with H.pylori infection (Positive for rapid urease test or 13C urea breath test).
3. Received at least two previous standard treatment protocols for Helicobacter pylori, and the application regimens included at least three low-resistance antibiotics.

Exclusion Criteria:

1. Patients with serious underlying diseases, such as liver insufficiency, renal insufficiency, immunosuppression, malignant tumors, Coronary heart disease or coronary artery stenosis ≥75%.
2. Patients who are pregnant or lactating or unwilling to take contraceptive measures during the trial.
3. Patients with active gastrointestinal bleeding.
4. Patients with a history of upper gastrointestinal surgery.
5. Patients allergic to treatment drugs.
6. Patients with medication history of bismuth agents, antibiotics, proton pump inhibitor and other drugs within 4 weeks
7. Patients with other behaviors that may increase the risk of illness, such as alcohol and drug abuse
8. Patients who are unwilling or incapable to provide informed consents.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study enrolled patients with extremely refractory Helicobacter pylori (H. pylori) infection, identified in the outpatient department. These patients had previously undergone eradication programs that included three antibiotics with low resistance rates: amoxicillin, tetracycline, and furazolidone. Despite this, reexamination confirmed persistent H. pylori infection. Upon entry into the study, participants were required to fulfill the inclusion criteria, not meet the exclusion criteria, and provide signed informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Eradication rate | Immediately after follow-up check.

SECONDARY OUTCOMES:
Rate of adverse reactions. | Immediately after follow-up check.
False positive rate | Immediately after follow-up check.
  The false positive rate is defined as the proportion of patients whose only C13 breath test results are positive and any other test is negative.
Patient compliance | Immediately after follow-up check.
  Good compliance is defined as the actual dosage is within the range of 80%-100% of the dosage that should be taken.
Cost-effectiveness index | Immediately after follow-up check.
  Ratio of costs to effectiveness

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided